CLINICAL TRIAL: NCT02890563
Title: Compression Therapy Following Truncal Vein Endothermal Ablation And Distal Sclerotherapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oulu University Hospital (Other)
Responsible Party: Principal Investigator, Toni Pihlaja, M.D., Oulu University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 131/2016
Record Dates: First submitted 2016-08-31; First posted 2016-09-07 (Estimated); Last update posted 2019-04-01 (Actual); Status verified 2019-03

CONDITIONS: Varicose Veins
Keywords: Varicose veins; Compression stockings; Sclerotherapy; Radiofrequency ablation
MeSH Terms: conditions — Varicose Veins

ARMS (2):
- No Compression (No Intervention): Patients in this group will not receive any compression after treatment.
- Compression (Active Comparator): Patients in this group will use compression stockings for seven days after treatment (2 days continuously and 5 days during daytime).
  Interventions: Device: Class II Compression Stockings

INTERVENTIONS:
Device: Class II Compression Stockings
  Arms: Compression

SUMMARY:
Study purpose is to research whether compression therapy is beneficial after truncal vein RF-ablation and distal sclerotherapy done in the same session when needed. Patients will be randomised to either no compression group (Group I) or compression group (Group II)

DETAILED DESCRIPTION:
In this study two endpoints are anticipated, first endpoint is to assess safety and adverse effects between groups at 1 month endpoint. Also post-procedural pain and need for painkillers are monitored. Compliance and reasons for non-compliance is recorded in compression group.

Second endpoint is to assess mid-term (6 months) success of truncal vein occlusion as well as changes in Aberdeen score between groups compared to pre-operative stage.

Study design is non-inferiority trial where in 5% margin occlusion of truncal vein is expected to be equal in two groups at 6 six months. Power analysis showed need for 85 patients per group and taking into account possible dropouts anticipated n = 200.

ELIGIBILITY:
Inclusion Criteria:

* Duplex ultrasound verified GSV and/or SSV incompetence (0.5 seconds or more)
* Comprehensive Classification System for Chronic Venous Disorders (CEAP) rated from C2 to C4
* Truncal vein insufficiency (GSV and/or SSV) treatable with Radiofrequency ablation

Exclusion Criteria:

* History of pulmonary embolism or deep venous thrombosis
* Large (>12mm) truncal vein diameter
* CEAP C5-C6
* Patient unwilling to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2016-08; Primary Completion 2019-03 (Actual); Study Completion 2019-03 (Actual)

PRIMARY OUTCOMES:
Truncal vein occlusion rate | 6 months

SECONDARY OUTCOMES:
Post-operative pain assessed with visual analogue scale (VAS) | 10 days
Painkillers usage after treatment | 10 days
  Need for Paracetamol/NSAIDs after treatment
Aberdeen Varicose Veins Questionnaire (AVVQ) | 6 months
  Assessed preoperatively and at one and six months
Compliance with compression stockings | 7 days
  To assess compliance and possible reasons for non-compliance at compression group
Time required returning to normal work and activity level | 14 days
Signs of deep venous thrombosis, pigmentation, blisters, skin irritation, thrombophlebitis, hematoma, wound infection or paraesthesia post operatively | 30days
  Assessed in 1month control and earlier if necessary (Patient is instructed to contact outpatient clinic in case of problems).

CONTACTS AND LOCATIONS:
Overall Officials: Toni Pihlaja, M.D., Principal Investigator — Oulu University Hospital
Locations (2):
- Finland (2):
  - Raahe's hospital, Raahe, North Ostrobothnia
  - Oulu University Hospital, Vascular Department, Oulu

REFERENCES:
- [Derived] Pihlaja T, Romsi P, Ohtonen P, Jounila J, Pokela M. Post-procedural Compression vs. No Compression After Radiofrequency Ablation and Concomitant Foam Sclerotherapy of Varicose Veins: A Randomised Controlled Non-inferiority Trial. Eur J Vasc Endovasc Surg. 2020 Jan;59(1):73-80. doi: 10.1016/j.ejvs.2019.08.020. Epub 2019 Nov 18. PMID 31753745